CLINICAL TRIAL: NCT07081126
Title: Daratumumab for Late Antibody-Mediated Rejection in Kidney Transplant Recipients With De Novo Donor-Specific Antibodies: A Case-Control Study
Brief Title: Daratumumab for Late Antibody-Mediated Rejection
Acronym: DARTABMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Matej Vnucak, MD, PhD, University Hospital, Martin
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TNO_UNM_DARA
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Kidney Tansplant; Acute Rejection (AR) of Transplanted Kidney
Keywords: daratumumab; kidney transplant; acute antibody mediated rejection
MeSH Terms: interventions — daratumumab; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dara (Active Comparator): Kidney transplant recipients with late ABMR and de novo DSA treated with daratumumab (1800mg subcutaneous, weekly x 4, then monthly x 6).
  Interventions: Drug: Daratumumab (Subcutaneously)
- control group (Other): Kidney transplant recipients with late ABMR and de novo DSA treated with standard therapies (IVIG, plasmapheresis, rituximab, etc.) prior to the start of the daratumumab study.
  Interventions: Other: control group

INTERVENTIONS:
Drug: Daratumumab (Subcutaneously) — Kidney transplant recipients with late ABMR and de novo DSA treated with daratumumab (1800mg subcutaneous, weekly x 4, then monthly x 6).
  Arms: Dara
Other: control group — Kidney transplant recipients with late ABMR and de novo DSA treated with standard therapies (IVIG, plasmapheresis, rituximab, etc.) prior to the start of the daratumumab study.
  Arms: control group

SUMMARY:
The study titled "Daratumumab for Late Antibody-Mediated Rejection in Kidney Transplant Recipients with De Novo Donor-Specific Antibodies" (DARTABMR) is a case-control investigation assessing whether daratumumab is more effective than standard therapies (such as IVIG, plasmapheresis, and rituximab) in treating late antibody-mediated rejection (ABMR) in kidney transplant patients with new donor-specific antibodies (DSA). The research compares outcomes like kidney function stabilization, DSA reduction, and biopsy improvements between patients receiving daratumumab and those on standard treatments. Participants include transplant recipients diagnosed with ABMR more than 12 months post-transplant, with data collected on clinical, immunological, and biopsy parameters before, during, and after treatment. The study emphasizes matching participants based on key variables to minimize bias and will analyze treatment success rates, changes in kidney function and DSA levels, and adverse events.

DETAILED DESCRIPTION:
The DARTABMR study is a comprehensive case-control research project designed to evaluate the efficacy of daratumumab in treating late antibody-mediated rejection (ABMR) in kidney transplant recipients with de novo donor-specific antibodies (DSA). The primary objective is to determine whether daratumumab offers superior outcomes compared to standard therapies like intravenous immunoglobulin (IVIG), plasmapheresis, and rituximab.

Study Design and Population:

This is a retrospective and prospective case-control study involving kidney transplant recipients diagnosed with late ABMR, defined as occurring more than 12 months post-transplant. Patients are divided into two groups: the case group receiving daratumumab (1800 mg subcutaneously, weekly for four doses, then monthly for six doses) and a control group previously treated with standard therapies. Inclusion criteria encompass first or subsequent kidney transplants with biopsy-proven ABMR and presence of de novo DSA. Exclusion criteria include active infections, significant comorbidities, prior daratumumab treatment, contraindications, and non-adherence to immunosuppression protocols. Patients are matched based on ABMR diagnosis timing, baseline kidney function, DSA characteristics, number of transplants, age, and ethnicity to minimize confounding.

Intervention and Data Collection:

All participants, both cases and controls, are maintained on a standardized immunosuppressive regimen consisting of tacrolimus, mycophenolate mofetil (MMF), and steroids, with specified targets and documentation of any deviations. Data collected encompass demographic information, clinical history, immunosuppressive details, kidney function tests (creatinine, eGFR), DSA levels (via Luminex), and biopsy findings using Banff scoring and molecular analyses. For the daratumumab group, assessments occur at baseline, during treatment, and after the last dose, including monitoring for infections, adverse events, and immune profiles via flow cytometry and cell-free DNA (cfDNA). For controls, retrospective data on treatment regimens, kidney function, DSA levels, biopsy results, infections, and safety are gathered.

Outcome Measures and Analysis:

The primary endpoint is treatment success, defined by improvement or stabilization of kidney function, significant reduction in DSA levels (e.g., ≥50% MFI decrease), and favorable biopsy changes. Graft survival during follow-up is also considered. Secondary analyses compare changes in kidney function, DSA levels, biopsy scores, and incidence of adverse events between groups. Statistical methods include chi-square or Fisher's exact tests for success rates, t-tests or ANOVA for continuous variables, and regression analyses to control for residual confounders.

Summary:

Overall, the DARTABMR aims to provide evidence on whether daratumumab can improve outcomes in late ABMR cases with de novo DSA, potentially influencing future treatment protocols for this challenging clinical scenario.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient (first or subsequent transplant)
* Diagnosis of late ABMR (diagnosed >12 months post-transplant)
* Biopsy-proven ABMR
* Presence of de novo DSA

Exclusion Criteria:

* Active infection
* Other significant comorbidities that could affect outcomes or treatment safety
* Contraindications to daratumumab
* Prior treatment with daratumumab
* Specific types of DSA (consider specifying, e.g., unacceptable antigens)
* Non-adherence to standardized immunosuppression protocol (tacrolimus, MMF, steroids)
* iFTA 2 or 3 on baseline biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Is daratumumab superior to standard therapies (IVIG, plasmapheresis, rituximab) in improving outcomes in kidney transplant recipients with late antibody-mediated rejection (ABMR) and de novo donor-specific antibodies (DSA)? | 7 months
  The primary outcome measure of the DARTABMR study is the proportion of kidney transplant recipients who achieve treatment success, defined by the following criteria:
  Improvement or stabilization of kidney function, indicated by no significant decline, or an increase in estimated glomerular filtration rate (eGFR).
  Reduction in donor-specific antibody (DSA) levels, with a clinically meaningful decrease, such as greater than 50% reduction in mean fluorescence intensity (MFI).
  Improvement in biopsy findings, evidenced by a reduction in Banff scores for features such as glomerulitis and peritubular capillaritis.
  The study will compare the percentage of patients meeting these criteria between the daratumumab-treated group and the standard therapy control group during the follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Martin, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT07081126/Prot_SAP_000.pdf